CLINICAL TRIAL: NCT05892276
Title: Effects of Cannabidiol on Memory Reconsolidation and Trauma-Related Symptoms: A Randomized Clinical Trial
Brief Title: Effects of CBD Oil on Memory Reconsolidation and Trauma-Related Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The UT IRB determined that CBD oil is being used as a drug as defined by the FDA. Therefore, an IND must be obtained for the use of CBD oil in this research study in accordance with FDA regulations, 21 CFR 312.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor of Clinical Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00004278
Record Dates: First submitted 2023-05-15; First posted 2023-06-07 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Cannabidiol; CBD; PTSD; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD-WR (Experimental): 300 mg CBD broad-spectrum oil will be administered within the reconsolidation window.
  Preclinical studies demonstrate that the disruptive effects of CBD oil on memory reconsolidation depend on the timing of pharmacological administration (within 6 hours of memory reactivation).
  Thus, participants will be asked to take a single 300mg oral dose of CBD broad-spectrum oil immediately after the trauma memory reactivation procedure.
  Interventions: Behavioral: Trauma Memory Reactivation; Dietary Supplement: Cannabidiol (CBD) Broad-Spectrum Oil
- PBO-WR (Placebo Comparator): Placebo oil will be administered within the reconsolidation window.
  Participants will be asked to take a single dose of an MCT coconut oil placebo solution immediately after the trauma memory reactivation procedure.
  Interventions: Behavioral: Trauma Memory Reactivation; Dietary Supplement: Placebo Oil
- CBD-OR (Active Comparator): 300mg CBD broad-spectrum oil will be administered outside of the reconsolidation window.
  Participants will be asked to take a single 300mg oral dose of CBD broad-spectrum oil approximately 24 hrs after the trauma memory reactivation procedure.
  Thus, CBD will be administered well beyond the critical period for memory reconsolidation. The inclusion of this third arm provides a more robust test of the specific reconsolidation theory-based study hypotheses and aids in controlling for any nonspecific possible anxiolytic effects of CBD.
  Interventions: Behavioral: Trauma Memory Reactivation; Dietary Supplement: Cannabidiol (CBD) Broad-Spectrum Oil

INTERVENTIONS:
Behavioral: Trauma Memory Reactivation — Participants will be guided through the trauma memory reactivation paradigm by the study staff. The trauma memory reactivation paradigm entails two distinct procedures: (1) participants will watch a video clip related to their trauma; then (2) describe a verbal narrative of their traumatic event for approximately 5 minutes to a research team member.
Dietary Supplement: Cannabidiol (CBD) Broad-Spectrum Oil — 300mg CBD broad-spectrum oil.
  Arms: CBD-OR; CBD-WR
Dietary Supplement: Placebo Oil — 3ml oral dose of medium-chain triglycerides (MCT) coconut oil.
  Arms: PBO-WR

SUMMARY:
The purpose of this study is to investigate the effects of cannabidiol (CBD) broad-spectrum oil on memory reconsolidation (memory storage) and trauma-related symptoms in trauma-exposed individuals after exposure to a trauma memory reactivation paradigm.

DETAILED DESCRIPTION:
It is estimated that over 70% of individuals worldwide have experienced a trauma during their lifetime. Many people spontaneously recover without formal intervention or treatment after exposure to a traumatic event; however, some individuals may develop intrusive trauma-related memories, avoidance, negative changes in cognition or mood, or changes in arousal and reactivity, resulting in clinical or subclinical symptoms of posttraumatic stress disorder (PTSD).

Recently, the potential therapeutic effects of cannabidiol (CBD) have been investigated as a treatment for physical and mental health issues. Preclinical trials with rodents suggest that CBD may disrupt the reconsolidation of conditioned fear memories when administered within the six-hour memory reconsolidation window. These preclinical findings suggest that CBD may be clinically useful for preventing or treating PTSD. Although promising, little translational research has investigated the disruptive effects of CBD on memory reconsolidation in a trauma-exposed human population.

The overarching objective of this study is to investigate the effects of CBD broad-spectrum oil on memory reconsolidation and trauma-related symptoms in trauma-exposed individuals after exposure to a trauma memory reactivation procedure. To accomplish this, participants will be randomized to one of three treatment conditions: (a) CBD oil administered within the reconsolidation window (CBD-WR), (b) placebo oil administered within the reconsolidation window (PBO-WR), or (c) CBD oil administered well outside of the accepted memory reconsolidation window (CBD-OR). Participants will undergo a trauma memory reactivation paradigm, rate their emotional distress level, and complete other trauma-related measures.

To the best of our knowledge, this is the first clinical trial to investigate the effects of CBD broad-spectrum oil on memory reconsolidation and trauma-related symptoms among trauma-exposed individuals following exposure to a trauma memory reactivation paradigm. Additionally, this proof-of-concept pilot trial aims to contribute to the development of a novel, brief, packageable, and cost-effective secondary prevention or treatment for individuals with trauma-related fear memories and symptoms of trauma.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 65;
* Fluent in written and spoken English;
* Has access to the internet;
* Access to a camera with video recording capability;
* History of trauma exposure to either a motor vehicle collision (MVC), sexual assault, physical assault, or combat;
* Willingness to refrain from all non-study cannabis use during the study period

Exclusion Criteria:

* Insufficient emotional reactivity to trauma video clips
* Presence of significant suicidality or a history of a suicide attempt within the past 6 months;
* History or current alcohol or substance use disorder within the past month;
* History of psychosis within the past 6 months;
* Changes in psychotropic medication (≤ 8 weeks);
* Currently receiving trauma-focused psychotherapy;
* Any medical problem that would preclude participation in the study (e.g., liver or renal abnormalities or disease);
* Any current medication that would preclude participation in the study (e.g., use of prescribed blood, such as warfarin; use of anti-seizure medications, such as valproate, lamotrigine, or clobazam; use of thyroid medications, such as levothyroxine; use of heart rhythm medications, such as amiodarone);
* Pregnant or planning to become pregnant within the next 6 weeks;
* Regular cannabis use;
* History of adverse reaction to CBD oil or other CBD products;
* Allergy to coconut or coconut oil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Momentary Assessment of Distress Scale | Change from Baseline to Two-week Follow-up
  The Momentary Assessment of Distress Scale (MADS) is a customizable sliding scale used to measure continuous real-time changes in levels of subjective emotional stress on scale from 0 (no distress) to 10 (extreme distress). The MADS is used to index changes in emotional reactivity during exposure to a trauma memory reactivation cue.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist | Change from Baseline to Two-week Follow-up
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) is a 20-item self-report questionnaire that assesses symptoms consistent with the DSM-5 diagnosis of PTSD. Respondents rate the frequency of each symptom over the last month utilizing a 5-point scale (0 indicating "not at all"; 4 indicating "extremely").
Posttraumatic Cognition Inventory | Change from Baseline to Two-week Follow-up
  The Brief Version of the Posttraumatic Cognitions Inventory (PTCI-9) is a 9-item questionnaire that assesses negative posttraumatic cognition. Items are rated on a 7-point Likert scale with 1 indicating "Totally disagree" and 7 indicating "Totally agree." The instrument consists of three subscales (self-blame, negative cognitions of the self, and negative cognitions of the world) to yield the total and subscale scores, with higher scores indicating more negative posttraumatic cognitions.
Posttraumatic Safety Behaviors Inventory | Change from Baseline to Two-week Follow-up
  The Posttraumatic Safety Behavior Inventory (PSBI) is a 13-item self-report questionnaire that assesses safety behaviors related to PTSD. Items are rated on a 5-point scale with 0 indicating "Never" and 4 indicating "Always." The first 10 items of the inventory yield a summed total score. The last three items of the inventory are open-ended to record safety behavior specific to the respondent and can be used in clinical applications. Higher scores suggest more engagement with PTSD safety behaviors.
Posttraumatic Growth Inventory | Change from Baseline to Two-week Follow-up
  The Posttraumatic Growth Inventory (PGTI) is a 21-item self-report scale that measures positive outcomes associated with traumatic events. Items are rated on a 6-point scale with 0 indicating "I did not experience this as a result of my crisis" and 5 indicating "I experienced this change to a very great degree as a result of my crisis." The inventory is comprised of five factors (appreciation of life relating to others, spiritual change, new possibilities, and personal strength).
Trauma Coping Self-Efficacy Scale | Change from Baseline to Two-week Follow-up
  The Trauma Coping Self-Efficacy (CSE-T) Scale - 9-item is a brief self-report scale that assesses perceptions of coping self-efficacy following a traumatic experience. Respondents rate their perceived capacity to handle demands related to their trauma on a 7-point scale (1 indicating "Not at all capable"; 7 indicating "Totally capable").
Connor-Davidson Resilience Scale | Change from Baseline to Two-week Follow-up
  The Connor-Davidson Resilience Scale - 10 item (CD-RISC-10) is a 10-item self-report questionnaire that assesses resilience (e.g., the ability to cope with adverse experiences). Respondents rate items utilizing a 5-point scale (0 indicating "not true at all"; 4 indicating "true nearly all the time"). The summation of all items yields a total score, ranging from 0 to 40, with higher scores suggesting greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- The Laboratory for the Study of Anxiety Disorders, The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Aguilar-Gaxiola S, Alonso J, Benjet C, Bromet EJ, Cardoso G, Degenhardt L, de Girolamo G, Dinolova RV, Ferry F, Florescu S, Gureje O, Haro JM, Huang Y, Karam EG, Kawakami N, Lee S, Lepine JP, Levinson D, Navarro-Mateu F, Pennell BE, Piazza M, Posada-Villa J, Scott KM, Stein DJ, Ten Have M, Torres Y, Viana MC, Petukhova MV, Sampson NA, Zaslavsky AM, Koenen KC. Trauma and PTSD in the WHO World Mental Health Surveys. Eur J Psychotraumatol. 2017 Oct 27;8(sup5):1353383. doi: 10.1080/20008198.2017.1353383. eCollection 2017. PMID 29075426
- [Background] Murkar A, Kent P, Cayer C, James J, Durst T, Merali Z. Cannabidiol and the Remainder of the Plant Extract Modulate the Effects of Delta9-Tetrahydrocannabinol on Fear Memory Reconsolidation. Front Behav Neurosci. 2019 Aug 1;13:174. doi: 10.3389/fnbeh.2019.00174. eCollection 2019. PMID 31417379
- [Background] Stern CAJ, de Carvalho CR, Bertoglio LJ, Takahashi RN. Effects of Cannabinoid Drugs on Aversive or Rewarding Drug-Associated Memory Extinction and Reconsolidation. Neuroscience. 2018 Feb 1;370:62-80. doi: 10.1016/j.neuroscience.2017.07.018. Epub 2017 Jul 17. PMID 28729064